CLINICAL TRIAL: NCT07398573
Title: Comparison of the Analgesic Efficacy of Caudal and Quadratus Lumborum Blocks With Pain Monitoring in Lower Abdominal Surgery in Children
Brief Title: Comparison of Caudal and Quadratus Lumborum Blocks With Pain Monitoring in Children
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, DILARA YIGIT, Sub-Investigator, Ankara Etlik City Hospital
Other Study IDs: AESH-EK-2025-225 03/09/2025
Record Dates: First submitted 2025-09-18; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Regional Anesthesia Success; Pain Monitor During Anesthesia; Quadratus Lumborum Nerve Block; Caudal Block for Postoperative Analgesia; Pediatric Anesthesia
Keywords: Pediatric Anesthesia; Regional Block; Pain Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- QUADRATUS LUMBORUM BLOCK GROUP: Intraoperatively, under ultrasound guidance, bilateral QL block with 0.5 ml/kg of 0.25% bupivacaine (maximum volume 20 ml) will be performed.
- CAUDAL BLOCK GROUP: Under ultrasound guidance, a caudal block with 1 ml/kg of 0.125% bupivacaine (maximum volume 20 ml) will be performed.

SUMMARY:
Study Type: Prospective, Randomized, Observational Clinical Study

Primary Purpose:

The primary objective of this study is to compare the analgesic efficacy of caudal block (CB) and quadratus lumborum block (QLB) in children undergoing lower abdominal surgery using objective pain monitoring methods.

Key Questions Addressed:

Does the quadratus lumborum block provide superior intraoperative and postoperative analgesia compared to the caudal block, as measured by the Pain Monitor (PAM) and the FLACC scale?

Is the PAM monitor a reliable tool for objectively assessing nociception and pain in children who are unable to verbally express pain?

Which regional anesthesia technique more effectively delays the time to first postoperative analgesic requirement and reduces total analgesic consumption?

Which method is associated with higher parental satisfaction and fewer postoperative side effects, such as postoperative nausea and vomiting?

Comparison Groups:

Children receiving ultrasound-guided quadratus lumborum block will be compared with those receiving caudal block.

Intervention Group:

Bilateral quadratus lumborum block with 0.5 mL/kg of 0.25% bupivacaine.

Active Comparator Group:

Caudal block with 1 mL/kg of 0.125% bupivacaine.

Participant Population:

A total of 68 children, aged 2 months to 6 years, with ASA physical status I-II, scheduled for elective lower abdominal surgeries (e.g., inguinal hernia repair, orchiopexy, hydrocele).

What Participants Will Do:

Participants will receive the assigned regional block as part of standard anesthetic care. Observational data will be collected as follows:

Intraoperative: Continuous nociception monitoring using the PAM device at predefined time points (during laryngeal mask airway insertion, block performance, surgical incision, 20 minutes after block performance, and extubation).

Postoperative: Pain assessment using the FLACC scale at 1, 2, and 4 hours in the post-anesthesia care unit.

Rescue analgesia (intravenous paracetamol) will be administered if the FLACC score is ≥4. Time to first analgesic administration and total analgesic consumption will be recorded.

Additional outcomes include postoperative nausea and vomiting (PONV) scores, Steward recovery scores, and parental satisfaction scores assessed using the Pediatric Parental Satisfaction Scale (PPPS).

Primary Outcome:

Intraoperative PAM index scores.

Secondary Outcomes:

Postoperative FLACC scores, time to first analgesic requirement, total postoperative analgesic consumption, incidence and severity of PONV, Steward recovery scores, and parental satisfaction (PPPS) scores.

DETAILED DESCRIPTION:
Study Title:

Comparison of the Analgesic Efficacy of Caudal and Quadratus Lumborum Blocks Using a Pain Monitor in Children Undergoing Lower Abdominal Surgery

Study Objectives

Primary Objective:

To compare the analgesic efficacy of caudal block and quadratus lumborum block (QLB) using an objective pain monitoring device (Pain Monitor; PAM).

Secondary Objectives:

To evaluate the postoperative analgesic efficacy of caudal block and QLB in lower abdominal surgeries.

To compare postoperative analgesia duration and analgesic requirements between the two groups.

To assess postoperative side effects associated with each regional anesthesia technique.

To evaluate postoperative parental satisfaction.

Materials and Methods

Children aged 2 months to 6 years with ASA physical status I-II, scheduled for elective lower abdominal surgeries (e.g., inguinal hernia repair, orchiopexy, hydrocele) performed by the pediatric surgery unit at Etlik City Hospital, will be included.

Participants will be randomized using the Research Randomizer program (https://www.randomizer.org/

) into either the caudal block group or the quadratus lumborum block group. A total of 68 participants will be enrolled, with 34 participants in each group.

Both regional anesthesia techniques and the use of the PAM device for intraoperative nociception monitoring are established components of standard clinical practice at the study institution. Therefore, all participants will receive these interventions as part of routine perioperative care, independent of study participation. The study design is prospective and observational, with no deviation from standard anesthetic management.

Demographic data, anesthesia duration, and surgical duration will be recorded. Written informed consent will be obtained from parents or legal guardians preoperatively.

Participants may receive routine oral premedication with midazolam (0.5 mg/kg) in the preoperative area. In the operating room, standard monitoring (SpO₂, ECG, non-invasive blood pressure) will be applied, followed by placement of the PAM monitor. A pediatric probe will be placed on the foot in children younger than 3 years, and an adult probe will be placed on the hand in children aged 3 years or older.

Standard anesthesia induction and maintenance will be performed (oxygen/air mixture, sevoflurane, propofol, laryngeal mask airway). Under ultrasound guidance, either a caudal block with 1 mL/kg of 0.125% bupivacaine (maximum 20 mL) or a bilateral quadratus lumborum block with 0.5 mL/kg of 0.25% bupivacaine (maximum 20 mL) will be administered.

Intraoperative PAM index values will be recorded at five predefined time points:

During laryngeal mask airway insertion

During block performance

At the first surgical incision

20 minutes after block performance

During extubation

Following emergence from anesthesia, the PAM monitor will be removed, and participants will be observed for up to 4 hours postoperatively.

Postoperative assessments will include:

FLACC pain scores

PONV scores

Steward recovery scores

Parental satisfaction scores (PPPS)

These assessments will be performed at 1, 2, and 4 hours postoperatively.

Rescue analgesia with intravenous paracetamol (15 mg/kg) will be administered if the FLACC score is ≥4, and the time to first administration will be recorded. Postoperative complications will also be documented.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients between 2 months and 6 years of age
2. Pediatric patients undergoing lower abdominal surgery
3. Family consent must be obtained
4. No contraindications to block (infection at the block site), coagulopathy (INR <1.4, platelets >100,000), local anesthetic allergy)
5. ASA I-II patients

Exclusion Criteria:

1. Severe systemic disease (ASA ≥III)
2. Infection at the block site
3. Coagulopathy (INR >1.4, platelets <100,000)
4. Local anesthetic allergy
5. Parental refusal
6. Children aged <2 months or >6 years

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 2 months to 6 years with ASA I-II status undergoing lower abdominal surgeries (e.g., inguinal hernia, orchiopexy, hydrocele) performed by the pediatric surgery unit at Etlik City Hospital will be included.
Sampling Method: Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Pain Index Scores Measured by MEDSTORM Pain Monitor (PAM) | Perioperative period, at the following predefined time points: At airway instrumentation (laryngeal mask airway insertion) During regional block performance At skin incision 20 minutes after block performance At emergence from anesthesia (extubation)
  The intraoperative analgesic efficacy of Caudal Block and Quadratus Lumborum (QL) Block will be assessed using the MEDSTORM Pain Monitor (PAM).
  The PAM provides a Pain Index score ranging from 0 to 10, reflecting the patient's nociceptive state and the need for analgesic intervention. Lower scores indicate better analgesic efficacy.
  Pain Index scores will be recorded at predefined perioperative time points. It is hypothesized that the QL block will result in lower intraoperative Pain Index scores compared to the caudal block.
  Pain Index interpretation:
  0-1: No additional analgesia required 2-3: Additional analgesia may be required 4-5: Additional analgesia is likely required 6-7: Additional analgesia is probably needed 8-10: Additional analgesia is required
  Perioperative period, at the following predefined time points:
  At airway instrumentation During regional block performance At skin incision 20 minutes after block performance At emergence from anesthesia

SECONDARY OUTCOMES:
Postoperative Pain Intensity Measured by FLACC Scale | Postoperative period, assessed at: 1 hour after surgery 2 hours after surgery 4 hours after surgery
  Postoperative pain intensity will be assessed using the FLACC behavioral pain scale in children undergoing lower abdominal surgery who receive either a Caudal Block or a Quadratus Lumborum (QL) Block.
  The FLACC scale evaluates five behavioral categories: Face, Legs, Activity, Cry, and Consolability.
  Each category is scored from 0 to 2, resulting in a total score ranging from 0 to 10, where higher scores indicate greater pain intensity.
Time to First Postoperative Analgesic Requirement | Postoperative period, up to 4 hours after surgery
  Outcome Measure Description
  The duration of postoperative analgesia will be assessed by recording the time from the end of surgery to the first requirement for rescue analgesia.
  The need for rescue analgesia will be determined based on postoperative pain assessment using the FLACC behavioral pain scale.
  A FLACC score ≥4 will be used as the predefined threshold for rescue analgesic administration.
  Unit of Measure Hours
Number of Participants Requiring Postoperative Rescue Analgesia | Postoperative period, assessed at: 1 hour 2 hours 4 hours after surgery
  Outcome Measure Description
  The requirement for postoperative rescue analgesia will be recorded based on FLACC pain scores assessed at predefined postoperative time points.
  Participants with a FLACC score ≥4 will be considered as requiring rescue analgesia according to the institutional postoperative analgesia protocol.
  Unit of Measure
  Number of participants
Total Postoperative Paracetamol Dose Administered | Time Frame Postoperative period, up to 4 hours after surgery
  Total postoperative rescue analgesic consumption will be recorded. Rescue analgesia will be administered intravenously as paracetamol at a dose of 15 mg/kg when the FLACC score is ≥4.
  The cumulative paracetamol dose administered during the postoperative observation period will be calculated for each participant.
  Unit of Measure
  mg/kg
Adverse Effects, Postoperative Nausea and Vomiting (PONV) Severity Score | Postoperative period, assessed at: 1 hour 2 hours 4 hours after surgery
  Postoperative nausea and vomiting (PONV) will be systematically evaluated using a standardized four-point ordinal scoring system to allow objective and consistent assessment of PONV severity in children receiving either a Caudal Block or a Quadratus Lumborum (QL) Block.
  PONV severity will be classified as follows:
  Score 0: No nausea or vomiting
  Score 1: Mild nausea or retching not requiring treatment
  Score 2: Moderate nausea or vomiting requiring rescue antiemetic therapy
  Score 3: Severe, persistent nausea or vomiting refractory to initial rescue therapy
  This scoring system enables quantitative comparison of PONV severity between the two regional anesthesia techniques.
  Unit of Measure
  PONV severity score (0-3)
Postoperative Parental Satisfaction Score Assessed by the Pediatric Parental Satisfaction Scale (PPPS) | Postoperative period, assessed at: 1 hour 2 hours 4 hours after surgery
  Postoperative parental satisfaction with perioperative anesthesia care will be evaluated using the Pediatric Parental Satisfaction Scale (PPPS), a validated questionnaire designed to quantitatively assess the satisfaction of parents or guardians of pediatric patients.
  The PPPS uses a 5-point Likert scale, which is converted into a numerical satisfaction score, with higher scores indicating greater satisfaction. The score is interpreted as follows:
  Score 1: Very dissatisfied
  Score 2: Dissatisfied
  Score 3: Neutral
  Score 4: Satisfied
  Score 5: Very satisfied
  This scale allows objective comparison of parental satisfaction between children receiving Caudal Block and Quadratus Lumborum (QL) Block.
  Unit of Measure
  PPPS score (1-5)
Postoperative Recovery Score Assessed by the Steward Score | Postoperative period, assessed at: 1 hour 2 hours 4 hours after surgery
  Outcome Measure Description
  Post-anesthetic recovery will be evaluated using the Steward Recovery Score, a standardized composite scoring system designed to provide a rapid and objective assessment of recovery following anesthesia in pediatric patients receiving either a Caudal Block or a Quadratus Lumborum (QL) Block.
  The Steward Score evaluates three domains:
  Consciousness (0-2)
  Airway (0-2)
  Motor activity (0-2)
  Each domain is scored from 0 to 2, resulting in a total score ranging from 0 to 6, with higher scores indicating better recovery status.
  A total Steward Score of 6 is generally considered to reflect adequate recovery and readiness for transfer from the Post-Anesthesia Care Unit (PACU).
  Unit of Measure
  Steward Recovery Score (0-6)

CONTACTS AND LOCATIONS:
Overall Officials: ASLI DONMEZ, Professor, Principal Investigator — Etlik City Hospital Health Science University
Locations (1):
- Etlik City Hospital, Ankara, YENIMAHALLE, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Because it was not specified in the ethics committee.

REFERENCES:
- [Background] Aksu C, Sen MC, Akay MA, Baydemir C, Gurkan Y. Erector Spinae Plane Block vs Quadratus Lumborum Block for pediatric lower abdominal surgery: A double blinded, prospective, and randomized trial. J Clin Anesth. 2019 Nov;57:24-28. doi: 10.1016/j.jclinane.2019.03.006. Epub 2019 Mar 6. PMID 30851499
- [Background] Ledowski T. Objective monitoring of nociception: a review of current commercial solutions. Br J Anaesth. 2019 Aug;123(2):e312-e321. doi: 10.1016/j.bja.2019.03.024. Epub 2019 Apr 30. PMID 31047645
- [Background] Zhu Y, Wu J, Qu S, Jiang P, Bohara C, Li Y. The analgesic effects of quadratus lumborum block versus caudal block for pediatric patients undergoing abdominal surgery: a systematic review and meta-analysis. Front Pediatr. 2025 Feb 6;13:1492876. doi: 10.3389/fped.2025.1492876. eCollection 2025. PMID 39981211
- See also: Quadratus lumborum block procedure guide — https://www.uptodate.com/contents/quadratus-lumborum-block-procedure-guide?search=quadratus%20lumborum%20block&source=search_result&selectedTitle=1~15&usage_type=default&display_rank=1

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-09-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT07398573/Prot_SAP_ICF_000.pdf